CLINICAL TRIAL: NCT06211348
Title: Genomic Sequencing in Anatomically Normal Fetuses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-38946
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Pregnant Individuals Requesting Standard Microarray

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Genomic Sequencing (Experimental)
  Interventions: Device: Genomic Sequencing

INTERVENTIONS:
Device: Genomic Sequencing — Individuals who request prenatal diagnostic testing with standard chromosomal microarray will be offered genomic sequencing (GS) as an option to assess for additional disease risk.

SUMMARY:
This cohort study will examine the clinical utility of genomic sequencing (GS) in patients undergoing prenatal diagnostic procedures (chorionic villus sampling or amniocentesis) for routine indications other than a structural fetal anomaly.

DETAILED DESCRIPTION:
Individuals who request prenatal diagnostic testing with standard chromosomal microarray will be offered GS as an option to assess for additional disease risk. The GS will be limited to evaluation of single gene disorders on a curated gene list developed by our multidisciplinary team of experts. This will include only pathogenic or likely pathogenic variants in genes associated with conditions with a well-defined phenotype that may include cognitive impairment or debilitating health conditions in childhood and/or conditions that will impact maternal, fetal, neonatal, or early childhood health management with significant perinatal or pediatric morbidity or mortality. GS test results will be reported to the research participant by a clinical geneticist or genetic counselor with expertise in exome sequencing. Participants may use this information for pregnancy management including termination of pregnancy. Participants will be offered analysis for secondary findings, as recommended by the American College of Medical Genetics and Genomics. Analysis and reporting of GS will be performed by the UCSF CLIA-certified Genomic Medicine Laboratory. Blood or saliva samples will be collected on both parents to allow trio GS to determine inheritance of any potentially significant fetal variants.

The project is exploratory in nature, with a goal of contributing to a growing body of evidence regarding the clinical utility of GS in the prenatal population.

ELIGIBILITY:
Inclusion Criteria:

Pregnant patients who are:

* Pregnant with a structurally normal fetus (singleton or multiple gestation)
* Planning to undergo prenatal diagnosis by either chorionic villus sampling or amniocentesis with chromosome microarray analysis for routine indications
* Planning, or have already completed expanded carrier screening

Exclusion Criteria:

Pregnant patients who:

* Decline prenatal diagnostic testing
* Are pregnant and their fetus has a known anomaly
* Declined chromosomal microarray analysis of expanded carrier screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Detection of pathogenic or likely pathogenic variants with genomic sequencing | Up to 2 months after enrollment
  Proportion of positive genetic diagnosis among all pregnancies with anatomically normal fetuses

CONTACTS AND LOCATIONS:
Overall Officials: Mary Norton, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No